CLINICAL TRIAL: NCT02721056
Title: A Phase I-II Study of NBTXR3 Activated by Sterostatic Body Radiation Therapy (SBRT) In the Treatment of Liver Cancers
Brief Title: NBTXR3 Crystalline Nanoparticles and Stereotactic Body Radiation Therapy in the Treatment of Liver Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The RP2D for intratumoral injection was determined. With the changing practice of medicine for HCC, it was decided to design an independent Phase II clinical study.
Sponsor: Nanobiotix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBTXR3-103
Record Dates: First submitted 2015-12-24; First posted 2016-03-28 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2020-10

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Dose escalation (volume) of NBTXR3 (SBRT 45 Gy [15 Gy x 3 fractions over 5 - 7 days] or 50 Gy [10 Gy x 5 fractions over 5 - 15 days]), to define the early dose limiting toxicities (DLTs) and the recommended dose (volume) for further development.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NBTXR3, IL or IA injection +SBRT (Experimental): * Patients will receive a single intralesional (IL) injection of NBTXR3 at four increasing dose levels (Volume levels) equivalent to: 10%, 15%, 22%, 33% and 42% of the baseline tumor volume, activated by SBRT.
  * Patients with primary and secondary nodular intra hepatic cancers only will receive a single superselective transcatheter arterial (IA) injection of NBTXR3 at five increasing dose levels (Volume levels) equivalent to: 10%, 15%, 22%, 33% and 45% of the baseline tumor volume, activated by SBRT.
  Interventions: Radiation: NBTXR3, IL or IA injection + SBRT

INTERVENTIONS:
Radiation: NBTXR3, IL or IA injection + SBRT — Patients will receive a single administration of NBTXR3 on day of injection, as intralesional or super selective transcatheter arterial injection activated by Stereotactic Body Radiation Therapy starting 24 hours post injection. The total radiotherapy dose will be 45 or 50 Gy, delivered as three fractions of 15 Gy or 5 fractions of 10 Gy each, over 5 to 15 days (45 or 50Gy, 15GyX3 or 10GyX5).

SUMMARY:
The purpose of this Phase I / II study is to evaluate the safety and preliminary efficacy of NBTXR3 nanoparticles given by intralesional (IL) or intraarterial (IA) injection and activated by Stereotactic Body Radiation Therapy in the treatment of liver cancers.

DETAILED DESCRIPTION:
PHASE I PART: Dose escalation and Recommended Dose (Volume) The purpose of the Phase I part of the study is to determine the Recommended Dose (volume), the safety profile and the feasibility of the treatment of NBTXR3 administered either by intrahepatic lesion injection or super selective transcatheter arterial injection and activated by stereotactic body radiation therapy (SBRT), in patients with liver cancers. Primary objective

- To determine the Recommended Dose(s) (volume(s)) and the early Dose Limiting Toxicity (DLT) of NBTXR3 administered either by intralesional injection or by super selective transcatheter arterial injection and activated by stereotactic body radiation therapy (SBRT) in patients with liver cancers

PHASE II PART: Safety and Efficacy evaluation Primary objectives

The primary objectives of the Phase II part are:

* To assess and characterize the safety profile, including liver function evaluation using MELD/MELD-Na and Child-Pugh scores, of NBTXR3 activated by SBRT, at the Recommended Dose(s)(Volume(s)) as determined previously in the Phase I part, in patients with liver cancers Clinical Investigation Plan - NBTXR3/103
* To evaluate the antitumor activity in terms of Complete Response Rate (CRR) of target lesions, as per mRECIST for HCC and RECIST version 1.1 for liver metastases at 12 weeks' post radiotherapy, of NBTXR3 activated by SBRT, at the Recommended Dose(s) (Volume(s)) as determined previously in the Phase I part, in patients with liver cancer.

ELIGIBILITY:
Secondary cancer, Liver metastases

Inclusion criteria:

* Age ≥ 18
* Written Informed Consent obtained, signed and dated
* ECOG performance status 0 or 1
* Life expectancy > 6 months
* Liver metastases from other primary cancers 1) with histologic confirmation of metastases, or 2) History of primary cancer with histology available and lesions in the liver consistent with metastases, or 3) histologic confirmation of primary cancer and a growing enhancing lesion in the liver consistent with a metastasis
* Unresectable tumor/s, based on the opinion of an experienced surgeon specializing in hepatic resection, or the patient must be medically inoperable
* Patients with extra-hepatic metastases controlled by supportive care or concomitant hormonotherapy are eligible.
* Previous liver resection or local treatment (radiofrequency ablative therapy, chemoembolization, microwave treatment…) is permitted
* Patients must have recovered from the effects of previous therapy (residual AE grade 0 or 1)
* Radiological disease progression according to the investigator evaluation or according to RECIST 1.1
* At least one tumor lesion that can be accurately measured in at least one dimension according to RECIST 1.1
* Normal permeability of hepatic artery evaluated by injected CT-scan (arterial phase)
* Total target volume of lesions < 500cc and < 50% of the total liver volume
* 700 cc of liver volume without tumor involvement and a radiation therapy dose < 15 Gy
* The following laboratory parameters:
* Platelet count ≥ 50 x 10^9/L
* Hemoglobin ≥ 8.5 g/dL
* Absolute neutrophil count ≥ 1.5 x 10^9/L,
* Prothrombin rate (PR)> 50%
* International Normalized Ratio (INR) < 1.5 or correctable with vitamin K. Patients receiving anti-coagulation or anti-aggregation therapy must stop temporarily during treatment.
* Total bilirubin <30 μmol/l
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x upper limit of normal
* Albumin >2.5 g/dL
* Very low or undetectable HBV DNA and HCV RNA
* Serum Creatinine ≤ 1.5 time the upper limit of normal value
* Glomerular Filtration Rate > 44mL/min/1.73m2
* All female patients of childbearing potential must have a negative serum/urinary pregnancy test within the 7 days prior to NBTXR3 administration. Otherwise, Patients must be post-menopausal, surgically sterile, or using 'effective contraception'. The definition of 'effective contraception' will be based on the judgment of the investigator.

Exclusion criteria:

* Patients with ongoing chronic active viral B or C hepatitis must have received an antiviral treatment with negative or very low viremia before the onset of the radiation therapy
* Biliary tract dilatation, biliodigestive anastomosis, bile duct drainage
* Uncontrolled extra-hepatic metastatic disease with a symptomatic treatment or well tolerated hormonotherapy (AE 0/1)
* Previous cancer cured for less than 2 years
* Previous anticancer treatment (chemotherapy or/and biologicals) with a wash out < 4 weeks
* Previous treatment with intra-arterial injection of Y90 loaded microspheres in the same hepatic lobe than the current tumor.
* Previous intra-arterial chemotherapy
* Prior radiation therapy to the right upper abdomen, precluding re-irradiation of the liver. That is, any previous radiation therapy in which a mean dose to the liver of 15 Gy in conventional fractionation was delivered, or previous doses to critical normal structures that would make re-irradiation unsafe
* Impossibility to follow the dosimetry constraints (mean total liver dose > 15Gy)
* Presence of arterio-venous intra tumoral shunting
* Encephalopathy related to liver failure
* Clinical ascitis
* Presence of another scalable tumor disease except cervical carcinoma in situ, treated basal cell carcinoma, or superficial bladder tumors (Ta, Tis &T1)
* Presence of hepato pulmonary syndrome
* Auto immune hemolytic anemia
* Auto immune disorder, excepted auto immune thyroiditis
* Uncontrolled hypertension or congestive heart failure
* Active coronary artery disease (myocardial infarction more than 6 months prior to study entry is permitted)
* Previous gastrointestinal bleed within the past 2 months
* Known syndrome AIDS-related illness or serious non controlled acute or chronic illness
* Active, clinically severe bacterial or fungal infections (> grade 2 NCI-CTCAE, version 5.0)
* Complete initial work up earlier than 4 weeks prior to patient registration
* Patient whose general health condition does not allow treatment feasibility
* Patients unable and/or unwilling to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Patients participating in another clinical investigation at the time of signature of the informed consent.

Primary cancer: Hepato Cellular Carcinoma - HCC

Inclusion criteria:

* Age ≥ 18
* Written Informed Consent obtained, signed and dated
* ECOG performance status 0 or 1
* Life expectancy > 3 months
* Histological or cytological diagnosis of Hepatocellular cancer or imaging diagnosis by the American Association for the Study of Liver Disease (AASLD) guidelines or European association for the Study of the Liver (EASL) guidelines.
* Patients with HCC:
* Without main branch or intrahepatic trunk portal vein tumor thrombosis (Vp3 or Vp4, respectively), with progression or recurrence of HCC after surgical or loco-regional treatment
* With main branch (right and/or left) or intrahepatic trunk portal vein tumor thrombosis (Vp3 or Vp4, respectively), AND without right atrial involvement.
* Recurrent intrahepatic cholangiocarcinoma is eligible only in the phase I part
* Liver cirrhosis Child Pugh A - B7
* Previous liver resection or local treatment (radiofrequency ablative therapy, chemoembolization, microwave treatment…) is permitted
* Patients with previous treatment with sorafenib or other targeted or systemic therapy are eligible if wash out > 4 weeks
* Patients must have recovered from the effects of previous therapy (residual AE grade 0 or 1)
* Radiological disease progression according to the investigator evaluation or according to RECIST 1.1
* At least one tumor lesion that can be accurately measured in at least one dimension according to RECIST 1.1
* Normal permeability of hepatic artery evaluated by injected CT-scan (arterial phase)
* Total target volume of lesions < 500cc and < 50% of the total liver volume
* 700 cc of liver volume without tumor involvement and a radiation therapy dose < 15 Gy
* The following laboratory parameters:
* Platelet count ≥ 50 x 10^9/L
* Hemoglobin ≥ 8.5 g/dL
* Absolute neutrophil count ≥ 1.5 x 10^9/L,
* Prothrombin rate (PR)> 50%
* International Normalized Ratio (INR) < 1.5 or correctable with vitamin K
* Patients receiving anti-coagulation or anti-agregant therapy must stop temporarily during treatment.
* Total bilirubin <30 μmol/l
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x upper limit of normal
* Albumin >2.5 g/dL
* Very low or undetectable HBV DNA and HCV RNA
* Serum Creatinine ≤ 1.5 time the upper limit of normal value
* Glomerular Filtration Rate > 44mL/min/1.73m2
* All female patients of childbearing potential must have a negative serum/urinary pregnancy test within the 7 days prior to NBTXR3 administration. Otherwise, Patients must be post-menopausal, surgically sterile, or using 'effective contraception'. The definition of 'effective contraception' will be based on the judgment of the investigator.

Exclusion criteria:

* Patient suitable for a curative treatment by surgery or local treatment (radiofrequency ablation, microwave treatment, etc.)
* Patients with ongoing chronic active viral B or C hepatitis, those patients must have received an antiviral treatment with negativation of the viremia or very low viremia before the onset of the radiation therapy
* Biliary tract dilatation, biliodigestive anastomosis, bile duct drainage
* Extrahepatic Portal Vein Tumor Thrombosis
* Extra-hepatic metastasis
* Previous cancer cured for less than 2 years
* Previous anticancer treatment (chemotherapy or/and biologicals) with a wash out < 4 weeks
* Previous treatment with intra-arterial injection of Y90 loaded microspheres in the same hepatic lobe than the current tumor.
* Previous intra-arterial chemotherapy
* Concurrent treatment with any other anticancer therapy, including chemotherapy, immunotherapy, targeted therapy, gene therapy, or patients planning to receive these treatments during the study. Hormonotherapy is permitted
* Prior radiation therapy to the right upper abdomen, precluding re-irradiation of the liver. That is, any previous radiation therapy in which a mean dose to the liver of 15 Gy in conventional fractionation was delivered, or previous doses to critical normal structures that would make re-irradiation unsafe
* Impossibility to follow the dosimetry constraints (mean total liver dose > 15Gy)
* Presence of arterio-venous intra tumoral shunting
* Encephalopathy related to liver failure
* Clinical ascitis
* Presence of another scalable tumor disease except cervical carcinoma in situ, treated basal cell carcinoma, or superficial bladder tumors (Ta, Tis &T1)
* Presence of hepato pulmonary syndrome
* Auto immune hemolytic anemia
* Auto immune disorder, excepted auto immune thyroiditis
* Uncontrolled hypertension or congestive heart failure
* Active coronary artery disease (myocardial infarction more than 6 months prior to study entry is permitted)
* Previous gastrointestinal bleed within the past 2 months
* Known syndrome AIDS-related illness or serious non- controlled acute or chronic illness
* Active, clinically severe bacterial or fungal infections (> grade 2 NCI-CTCAE, version 5.0)
* Complete initial work up earlier than 4 weeks prior to patient registration
* Patient whose general health condition does not allow treatment feasibility
* Patients unable and/or unwilling to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* Patients participating in another clinical investigation at the time of signature of the informed consent. Phase I and II parts target the same liver cancer populations (same inclusion and

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-06 (Actual)

PRIMARY OUTCOMES:
Determination of the Recommended Doses Toxicities (DLT) | 50 Months
  To determine the Recommended Doses (DLT) of NBTXR3 administered as two different schedules (intra-lesional or intra-arterial injection), activated by Stereotactic Body Radiation Therapy (SBRT)
Determination of the early Dose Limiting Toxicities | 50 Months
  To determine the early Dose Limiting Toxicities

SECONDARY OUTCOMES:
Number of patients with treatment-related adverse events as assessed by CTCAE v4.0 | 50 Months
Response Rate | 50 Months
  To evaluate the antitumor activity in terms of Response Rate (RR) of target lesions/s, as per mRECIST and RECIST 1.1 criteria
Local Progression Free Survival | 50 Months
  To evaluate the local control in terms of local Progression Free Survival

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU La Croix Rousse, Lyon
  - Institut de Cancérologie de Loraine, Nancy
  - CHU de NANCY, Nancy
  - Centre René Gauducheau, Nantes
  - Hôpital Haut-Lévêque, Pessac
  - Centre Eugène Marquis, Rennes
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No